CLINICAL TRIAL: NCT05744544
Title: Sensory Assessment and Regression Rate of Bilateral External Oblique Intercostal Block and m-TAPA Block in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Sensory Assessment and Regression Rate of Bilateral External Oblique Intercostal Block and m-TAPA Block
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: DERMATOM55
Record Dates: First submitted 2023-01-16; First posted 2023-02-27 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Pain, Postoperative; Pain, Acute; Pain
Keywords: cutaneous block; Sensory Assessment; Regression Rate
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- External Oblique Intercostal Block Group: Sensory Assessment and Regression Rate will be performed on the anterolateral abdominal wall after EOIB. (external oblique intercostal block)
  Interventions: Procedure: External Oblique Block
- modified-TAPA block: Sensory Assessment and Regression Rate will be performed on the anterolateral abdominal wall after m-Tapa. (modified- thoracoabdominal nerves block through perichondrial approach)
  Interventions: Procedure: m-TAPA block

INTERVENTIONS:
Procedure: External Oblique Block — Patients will be followed after EOIB which are routinely performed in our clinic.
  Groups: External Oblique Intercostal Block Group
Procedure: m-TAPA block — m-TAPA block
  Groups: modified-TAPA block

SUMMARY:
External oblique and m-tapa blocks are routinely performed on patients undergoing laparoscopic cholecystectomy in our clinic. In this study, sensory block and regression rates will be investigated in patients who underwent block.

DETAILED DESCRIPTION:
External oblique block and m-Tapa blocks may be the key to provide adequate analgesia in patients undergoing abdominal surgery by blocking the abdominal nerves. In this study, the sensory dermatome block area calculation and the regression rate of the blocks will be evaluated in patients who underwent EOIB and m-Tapa.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing L/S cholecystectomy

Exclusion Criteria:

* patients who do not want to participate

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing L/S cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Sensory Assessment on the anterolateral abdominal wall | 24 hours
  Sensory Assessment will be performed on patients following the block procedure with pinprick test.
Regression Rate of the cutaneous block on anterolateral abdominal wall | 24 hours
  Regression Rate will be performed on patients following the block procedure with pinprick test.

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Tulgar, M.D., Study Chair — Samsun University
Locations (1):
- Samsun University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chen Y, Shi K, Xia Y, Zhang X, Papadimos TJ, Xu X, Wang Q. Sensory Assessment and Regression Rate of Bilateral Oblique Subcostal Transversus Abdominis Plane Block in Volunteers. Reg Anesth Pain Med. 2018 Feb;43(2):174-179. doi: 10.1097/AAP.0000000000000715. PMID 29278604
- [Result] Stoving K, Rothe C, Rosenstock CV, Aasvang EK, Lundstrom LH, Lange KH. Cutaneous Sensory Block Area, Muscle-Relaxing Effect, and Block Duration of the Transversus Abdominis Plane Block: A Randomized, Blinded, and Placebo-Controlled Study in Healthy Volunteers. Reg Anesth Pain Med. 2015 Jul-Aug;40(4):355-62. doi: 10.1097/AAP.0000000000000252. PMID 25923818